CLINICAL TRIAL: NCT02866786
Title: The Effects of Treatment With Oral Contraceptive Pill Containing Ethinyl Estradiol-Cyproterone Acetate and Metformin on Clinical, Hormonal, Metabolic and Ultrasonographic Characteristics in Polycystic Ovarian Syndrome
Brief Title: The Effects of OCP and Metformin on Clinical, Hormonal, Metabolic and Ultrasonographic Characteristics in PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: S.C.B. Medical College and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OG/2016/13
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Cyproterone acetate, ethinyl estradiol drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OCP only arm (Active Comparator): OCP containing 35 microgram ethinyl estradiol and 2 milligram cyproterone acetate to taken from the first day of the menstruation, oral administration of one pill daily for 21 days consecutively, then discontinue using the pill for seven days, and on the eighth day, restart taking the pill. OCP to be taken for 6 months.
  Interventions: Drug: ethinyl estradiol and cyproterone acetate
- Metformin arm (Active Comparator): Metformin 500mg bid in morning and evening after meals to be taken for 6 months.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin
  Arms: Metformin arm
Drug: ethinyl estradiol and cyproterone acetate — Oral Contraceptive Pill
  Arms: OCP only arm

SUMMARY:
Polycystic ovary syndrome (PCOS) is one of the most common endocrine disorder in women of reproductive age and is a leading cause of infertility due to anovulation. Oral contraceptive pills (OCPs) are considered as first line medical therapy to regularize menses in woman with PCOS. However they may worsen the metabolic profile of patients by elevating insulin resistance which is already deranged in PCOS. As there is higher prevalence of insulin resistance in Indian women with PCOS, insulin sensitisers like metformin may be more beneficial. Hence this study is undertaken to compare the combined effect of metformin and OCPs on the clinical, hormonal, metabolic and ovarian ultrasonographic characteristics in patients with PCOS and to evaluate whether this combination of drugs is more advantageous than OCPs or metformin alone in improving the clinical and metabolic profile.

DETAILED DESCRIPTION:
We aim to enroll about 120 patients fulfilling the Rotterdam diagnostic criteria for PCOS in our study. Patients will have a baseline clinical examination (Body weight, Body mass index, Waist circumference, Hirsutism score), hormonal profile (FSH, LH, fasting Insulin/glucose ratio, DHEAS, testosterone levels), metabolic profile (fasting and 2 hour post prandial plasma glucose, total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides level), ultrasound examination (ovarian volume and subcapsular follicle count, stromal echogenicity) and doppler blood flow study (ovarian stromal velocity, Pulsatility index, Resistivity index, Systolic/Diastolic ratio and stromal vascularization index).

Patients will be then randomized using a computer generated randomization program into two groups according to BMI (<25 and >25). The randomization will be stratified in order to achieve a homogenous distribution of PCOS patients in both arms of the study with respect to age and body mass index. Each group will be further subdivided into three treatment arms. 1st treatment arm will receive OCP containing 35 microgram ethinyl estradiol and 2 mg cyproterone acetate cyclically (21 days regimen) daily; 2nd treatment arm will receive OCP containing 35 microgram ethinyl estradiol and 2 mg cyproterone acetate cyclically (21 days regimen) while the 3rd treatment arm will receive OCP plus metformin 500 mg twice daily for a period of six months. Each patient will be asked to keep a diary of her menstrual periods over the study period. The patients will be followed up at 3 and 6 months of treatment to evaluate the changes in the above mentioned parameters. Analysis of the data will be done through descriptive and perceptive statistical methods by using Statistical Package for the Social Sciences (SPSS) software.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included into study who fulfill the Rotterdam diagnostic criteria (2003) for PCOS.

Exclusion Criteria:

* Current or previous use of oral contraceptives, glucocorticoids, antiandrogens, ovulation induction agents, antidiabetic and anti-obesity drugs or other hormonal drugs.
* Medical or surgical treatment of PCOS during the previous 3 months
* Presence of other endocrinopathies; except treated hypothyroidism on stable replacement doses of thyroid hormone
* Pregnancy, breastfeeding or desire for pregnancy during study interval (6 months)
* Inability to understand the proposal of the study precluding effective informed consent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Improvement in menstrual cycle pattern | 6 months
  All the participants will be asked to maintain a menstrual calendar and fill a questionnaire before and at the end of study. The questionnaire will include menstrual cycle dates, duration and amount from which improvement of menstrual pattern will be assessed.
Change in Abdominal Fat as measured by Waist Circumference in centimeter | 6 months
Change in weight as measured in kg | 6 months
Improvement in hirsutism measured by Modified Ferriman and Gallwey scores | 6 months
Improvement in glucose tolerance (measured by of fasting plasma glucose and 2-hour post prandial plasma glucose) | 6 months
Change in waist-to-hip ratio | 6 months
Change in Body mass index (kg/m2) | 6 months

SECONDARY OUTCOMES:
Lipid profile (Cholesterol, LDL, HDL and Triglyceride) improvement | 6 months
  The serum levels of Cholesterol, LDL, HDL and Triglyceride were measured in mg/dl before and after of treatment in both groups.
Change in blood level of luteinizing hormone [LH] (mIU/ml) | 6 months
Change in blood level of follicle stimulating hormone [FSH] (mIU/ml) | 6 months
Change in blood level of Testosterone (nmol/L) | 6 months
Change in blood level of Sex hormone binding globulin (SHBG) (ng/ml) | 6 months
Change in Free androgen Index (FAI) | 6 months
  Free Androgen Index or FAI is a ratio used to determine abnormal androgen status. The ratio is the total testosterone level divided by the sex hormone binding globulin (SHBG) level, and then multiplying by 100.
Change in Dehydroepiandrosterone sulfate (DHEAS) level (microgram/dl) | 6 months
Changes in fasting serum insulin levels (mIU/L) | 6 months
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | 6 months
  Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin concentrations. HOMA-IR = (Glucose x Insulin) / 405; Glucose is expressed in mg/dl and Insulin is expressed in mIU/L
Ovarian Stromal artery Pulsatility index | 6 months
Ovarian Stromal artery Resistivity index | 6 months
Chang in ovarian Follicle number by Ultrasonography (USG) | 6 months
  Largest cross-sectional plane of the ovary will be evaluated for follicle number
Change in ovarian Follicle diameter (in mm) by USG | 6 months
  Largest cross-sectional plane of the ovary will be evaluated for follicle diameter
Change in Ovarian volume (in cc) by USG | 6 months
  Ovarian volume, estimated according to the formula 1/2 (A x B x C), where A is the longitudinal diameter, B the anteroposterior diameter, and C the transverse diameter of the ovary
Change in Endometrial thickness (in mm) | 6 months
Change in ovarian stromal/total area ratio (S/A) | 6 months
  Ovarian area, evaluated by outlining with the caliper the external limits of the ovary in the maximum plane section. Ovarian stromal area, evaluated by outlining with the caliper the peripheral profile of the stroma, identified by a central area slightly hyperechoic with respect to the other ovarian area.

CONTACTS AND LOCATIONS:
Overall Officials: Mahija Sahu, MD, Principal Investigator — S.C.B. Medical College and Hospital; Priyadarshini Tripathy, MD, Principal Investigator — S.C.B. Medical College and Hospital
Locations (1):
- Department of Obstetrics & Gynecology, Cuttack, Odisha, India

IPD SHARING:
Plan to Share IPD: Yes